CLINICAL TRIAL: NCT06962943
Title: The Additional Effect of Auto-Regulated Blood Flow Restriction Exercise on Functional Performance and Muscle Fatigability in Athletes With Recurrent Ankle Sprain: A Randomized Controlled Clinical Study
Brief Title: Auto-regulated Blood Flow Restriction in Athletes With Recurrent Ankle Sprain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Prince Sattam Bin Abdulaziz University (Other)
Collaborators: University of Sharjah (Other)
Responsible Party: Principal Investigator, Walid Kamal Abdelbasset, PhD, Professor, Prince Sattam Bin Abdulaziz University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC-23-08-28-02-PG; University of Sharjah (Other: University of Sharjah)
Record Dates: First submitted 2025-04-30; First posted 2025-05-08 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Ankle Sprain; Ankle Instability
Keywords: Ankle instability; Blood flow restriction; Fatigability
MeSH Terms: conditions — Ankle Injuries | interventions — Control Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Auto-regulated blood flow restriction training (ARBFRT+TT) (Experimental): This group was recruited to conduct auto-regulated blood flow restriction exercise for 30-min, three times a week for six weeks by a trained physiotherapist.
  Interventions: Other: Auto-regulated Blood Flow Restriction Training
- Non-regulated blood flow restriction training (NRBFRT+TT) (Active Comparator): This group was recruited to conduct non-regulated blood flow restriction exercise for 30-min, three times a week for six weeks by a trained physiotherapist.
  Interventions: Other: Non-regulated Blood Flow Restriction Training
- Control group (Placebo Comparator): The control group was recruited to conduct no blood flow restriction exercise (Cuff with 0 pressure) 30-min, three times a week for 6 weeks.
  Interventions: Other: Control group

INTERVENTIONS:
Other: Auto-regulated Blood Flow Restriction Training — This group was recruited to conduct auto-regulated blood flow restriction exercise for 30-min, three times a week for six weeks by a trained physiotherapist, the subjects were asked to perform the following exercises: standing single leg calf raises with lateral resistance using a band, seated soleus raise, single leg balance on the edge of a step clearing the front foot with band on the big toe. SmartCuff 3.0 BFRT tool was used to automatically determine the individualized 50% arterial blood occlusion pressure for the BFRT group at the femoral artery, the cuff was connected to the smart tool device for the auto-regulated group to regulate the cuff pressure during muscle contraction and relaxation. The cuff was deflated in between exercises.
  Arms: Auto-regulated blood flow restriction training (ARBFRT+TT)
Other: Non-regulated Blood Flow Restriction Training — This group was recruited to conduct a non-regulated blood flow restriction exercise for 30-min, three times a week for six weeks by a trained physiotherapist, the subjects were asked to perform the following exercises: standing single leg calf raises with lateral resistance using a band, seated soleus raise, single leg balance on the edge of a step clearing the front foot with band on the big toe. SmartCuff 3.0 BFRT tool was used, whilst the cuff was not connected to the device in the non-regulated blood flow restriction training group and the pressure was stabilized as the initial pressure determined by the device in the non-regulated group. The cuff was deflated in between exercises.
  Arms: Non-regulated blood flow restriction training (NRBFRT+TT)
Other: Control group — This group was recruited to conduct no blood flow restriction exercise 30 min, three times a week for 6 weeks. SmartCuff 3.0 BFRT tool was used, whilst the cuff was not connected to the device and the pressure was 0 (zero) in this group. The cuff was deflated in between exercises.
  Arms: Control group

SUMMARY:
Ankle injuries, especially lateral ankle sprains, are prevalent in physically active individuals. Blood Flow Restriction Training (BFRT) has emerged as a promising method, employing partial arterial occlusion and full venous occlusion with low resistance to induce metabolic stress and achieve outcomes akin to heavy resistance training. This Randomized Controlled study explores the application of BFRT in addressing Chronic Ankle Instability (CAI), focusing on its efficacy in strength gains of extrinsic foot muscles, and potential benefits in functional performance.

DETAILED DESCRIPTION:
Ankle injuries, especially lateral ankle sprains, are prevalent in physically active individuals. Blood Flow Restriction Training (BFRT) has emerged as a promising method, employing partial arterial occlusion and full venous occlusion with low resistance to induce metabolic stress and achieve outcomes akin to heavy resistance training.

This Randomized Controlled study explores the application of BFRT in addressing Chronic Ankle Instability (CAI), focusing on its efficacy in strength gains of extrinsic foot muscles, and potential benefits in functional performance.

At the Sharjah University Medical Campus, 45 athletes from Shabab Al Ahli Club, aged 18-40, participated in this randomized control study. The investigators randomly allocated the participants into three equal groups, with 15 individuals in each group. The investigators recruited the first group to an auto-regulated blood flow restriction training plus traditional treatment program (ARBFRT+TT), the second group to a non-regulated blood flow restriction training plus traditional treatment program (NRBFRT+TT), and the third group to a traditional treatment program only without BFRT (TT group). The investigators assessed extrinsic foot muscle strength using an isokinetic device and functional performance using Functional Ankle Disability Index (FADI) and Rate of perceived exertion scale (RPES), both pre- and post 6-week treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age ranges from 18 to 40 years.
* No other health related conditions such as diabetes or hypertension.
* Unilateral or bilateral CIA.
* Male Athletes.

Exclusion Criteria:

* Knee or hip injury within the last 3 months.
* Previous ankle surgery.
* Any contraindication for BFRT application such as venous insufficiency, arterial insufficiency, history of DVT.
* Spinal lesion affecting lower limb function.
* Females

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-01-30 (Actual); Study Completion 2024-02-02 (Actual)

PRIMARY OUTCOMES:
Muscle Strength | 6 weeks
  An isokinetic dynamometer (Physiomed Elektromedizin AG [TP Module, CON-TREX MJ], Schnaittach, Germany) was used for strength testing. Using the previously identified ankle evertors/invertors and plantarflexors/dorsiflexors muscles, the investigators assessed the average peak torque to body weight ratio (concentric/concentric) at an angular velocity of 60°/s. Calibration of the dynamometer was performed prior to evaluation. Submaximal three and maximal three exercise sessions were given to participants to acclimate them to the testing methodology. Each subject rested for two minutes before cycling through the active range of motion three times in a row at maximum concentric contraction. To provide sufficient recovery between contractions, a 5-minute rest interval was included in each test condition. It was expected that participants would give it their all when taking the exam. For every test, the appropriate ankle isokinetic device was used for strength testing.

SECONDARY OUTCOMES:
Foot and ankle disability index | 6 weeks
  For the purpose of clinical treatment and research investigations involving young people with chronic ankle instability, the foot and ankle disability index (FADI) self-report measure was advocated. Results showed that it was responsive, reliable, and valid for patients with chronic ankle instability. There are a total of 26 items: 22 that pertain to activities and 4 that are associated with pain. The activity item is assessed on a scale from 0 (very difficult) to 4 (very easy), whereas the FADI 4 pain items are graded from 0 (very terrible pain) to 4 (very little pain) (Hale and Hertel, 2005). The overall value of the FADI is 104 points. A score of 100% on the FADI indicated that there was no abnormality.
Fatigability level | 6 weeks
  The Rating of Perceived Exertion scale (RPES) was used to assess the level of fatigability, which ranges from 0 to 10, was used to describe the amount of exhaustion experienced by the participants just before to their injuries. A score of 0 indicates that there was no effort at all, while a score of 10 indicates that the exertion was exceedingly intense. The quantity of typical physical activity, measured in hours per week, that was performed, was recorded in order to ascertain the degree of physical fitness achieved

CONTACTS AND LOCATIONS:
Overall Officials: Abdelbasset, Principal Investigator — University of Sharjah
Locations (1):
- Walid Kamal Abdelbasset, Sharjah city, Emirate of Sharjah, United Arab Emirates